CLINICAL TRIAL: NCT02482610
Title: Regulation of Postprandial Nitric Oxide Bioavailability and Vascular Function By Dairy Fat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Richard Bruno, Professor and Principal Investigator, Ohio State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2015H0088B
Record Dates: First submitted 2015-06-24; First posted 2015-06-26 (Estimated); Results first posted 2019-04-29 (Actual); Last update posted 2019-04-29 (Actual); Status verified 2019-04

CONDITIONS: Prediabetes
Keywords: Dairy; Milk; Glucose; Postprandial; Hyperglycemia; Prediabetes; Blood glucose; Oxidative stress; Vascular health; Vascular function
MeSH Terms: conditions — Prediabetic State; Hyperglycemia | interventions — Glucose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Glucose (Active Comparator): This study day will last approximately three hours and will be separated from the other arms by four days for men and one month for women.
  Interventions: Other: Glucose
- Glucose with Whole Fat Milk (Experimental): This study day will last approximately three hours and will be separated from the other arms by four days for men and one month for women.
  Interventions: Other: Glucose with Whole Fat Milk
- Glucose with Non-fat Milk (Experimental): This study day will last approximately three hours and will be separated from the other arms by four days for men and one month for women.
  Interventions: Other: Glucose with Non-fat Milk

INTERVENTIONS:
Other: Glucose — Following baseline measurements, participants will consume a 75 g glucose solution within five minutes.
  Arms: Glucose
Other: Glucose with Whole Fat Milk — Following baseline measurements, participants will consume 75 g glucose dissolved in two cups of whole fat milk within five minutes.
  Arms: Glucose with Whole Fat Milk
Other: Glucose with Non-fat Milk — Following baseline measurements, participants will consume 75 g glucose dissolved in two cups of non-fat milk within five minutes.
  Arms: Glucose with Non-fat Milk

SUMMARY:
Cardiovascular disease (CVD) is the leading cause of death in the United States. Short-term increases in blood sugar, or postprandial hyperglycemia (PPH), affect blood vessel function and increase the risk of CVD. Greater intakes of dairy foods have been associated with a lower risk of CVD, but whether these effects occur directly or indirectly by displacing foods in the diet that might increase CVD risk is unclear. Further controversial is the extent to which dietary fat derived from dairy foods regulate the risk of CVD. The health benefits of dairy on CVD risk are at least partly attributed to its ability to limit PPH and resulting PPH-mediated responses leading to vascular dysfunction. This provides rationale to investigate full-fat containing dairy as a dietary strategy to reduce PPH and risk for heart disease. The objective of this project is to define the extent to which full-fat dairy milk compared to non-fat dairy milk protects against PPH-induced vascular dysfunction by reducing oxidative stress responses that limit nitric oxide bioavailability to the vascular endothelium in adults with prediabetes.

DETAILED DESCRIPTION:
This study consists of three, 3-hour postprandial trials in response to consuming the following dietary treatments: 1. oral glucose challenge, 2. oral glucose challenge in combination with non-fat milk, and 3. oral glucose challenge in combination with whole milk. For three days preceding each trial, participants will be provided all meals to standardize physiologic responses to test meals. On each trial day, vascular function will be assessed and blood samples collected prior to and at 30 minute intervals for 3 hours following test meal ingestion.

ELIGIBILITY:
Inclusion Criteria:

1. hemoglobin A1c 5.7-6.4%
2. non-dietary supplement user
3. no medications affecting vasodilation, inflammation, or energy metabolism
4. no CVD
5. nonsmokers
6. individuals having blood pressure <140/90 mmHg and total cholesterol <240 mg/dL

Exclusion Criteria:

1. unstable weight (±2 kg)
2. vegetarian or dairy allergy
3. alcohol intake >3 drinks/day or >10 drinks/week
4. ≥ 7 hours/week of aerobic activity

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2018-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard S Bruno, PhD, RD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

REFERENCES:
- [Background] Mozaffarian D, Benjamin EJ, Go AS, Arnett DK, Blaha MJ, Cushman M, de Ferranti S, Despres JP, Fullerton HJ, Howard VJ, Huffman MD, Judd SE, Kissela BM, Lackland DT, Lichtman JH, Lisabeth LD, Liu S, Mackey RH, Matchar DB, McGuire DK, Mohler ER 3rd, Moy CS, Muntner P, Mussolino ME, Nasir K, Neumar RW, Nichol G, Palaniappan L, Pandey DK, Reeves MJ, Rodriguez CJ, Sorlie PD, Stein J, Towfighi A, Turan TN, Virani SS, Willey JZ, Woo D, Yeh RW, Turner MB; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2015 update: a report from the American Heart Association. Circulation. 2015 Jan 27;131(4):e29-322. doi: 10.1161/CIR.0000000000000152. Epub 2014 Dec 17. No abstract available. PMID 25520374
- [Background] DECODE Study Group, the European Diabetes Epidemiology Group.. Glucose tolerance and cardiovascular mortality: comparison of fasting and 2-hour diagnostic criteria. Arch Intern Med. 2001 Feb 12;161(3):397-405. doi: 10.1001/archinte.161.3.397. PMID 11176766
- [Background] Ballard KD, Bruno RS. Protective role of dairy and its constituents on vascular function independent of blood pressure-lowering activities. Nutr Rev. 2015 Jan;73(1):36-50. doi: 10.1093/nutrit/nuu013. PMID 26024056
- [Background] Ballard KD, Mah E, Guo Y, Pei R, Volek JS, Bruno RS. Low-fat milk ingestion prevents postprandial hyperglycemia-mediated impairments in vascular endothelial function in obese individuals with metabolic syndrome. J Nutr. 2013 Oct;143(10):1602-10. doi: 10.3945/jn.113.179465. Epub 2013 Aug 21. PMID 23966328
- [Result] McDonald JD, Mah E, Chitchumroonchokchai C, Dey P, Labyk AN, Villamena FA, Volek JS, Bruno RS. Dairy milk proteins attenuate hyperglycemia-induced impairments in vascular endothelial function in adults with prediabetes by limiting increases in glycemia and oxidative stress that reduce nitric oxide bioavailability. J Nutr Biochem. 2019 Jan;63:165-176. doi: 10.1016/j.jnutbio.2018.09.018. Epub 2018 Sep 25. PMID 30412905

RESULTS

PARTICIPANT FLOW:
Groups:
- Glucose, Then Glucose +Non-fat Milk, Then Glucose + Whole Milk: Each study day lasted approximately three hours and was separated from the other arms by four days for men and one month for women.
  Glucose: Following baseline measurements, participants consumed a 75 g glucose solution within five minutes.
  Glucose with Non-fat Milk: Following baseline measurements, participants consumed 75 g glucose dissolved in two cups of non-fat milk within five minutes.
  Glucose with Whole Fat Milk: Following baseline measurements, participants consumed 75 g glucose dissolved in two cups of whole fat milk within five minutes.
- Glucose, Then Glucose + Whole Milk, Then Glucose +Non-fat Milk: Each study day lasted approximately three hours and was separated from the other arms by four days for men and one month for women.
  Glucose: Following baseline measurements, participants consumed a 75 g glucose solution within five minutes.
  Glucose with Whole Fat Milk: Following baseline measurements, participants consumed 75 g glucose dissolved in two cups of whole fat milk within five minutes.
  Glucose with Non-fat Milk: Following baseline measurements, participants consumed 75 g glucose dissolved in two cups of non-fat milk within five minutes.
- Glucose +Non-fat Milk, Then Glucose + Whole Milk, Then Glucose: Each study day lasted approximately three hours and was separated from the other arms by four days for men and one month for women.
  Glucose with Non-fat Milk: Following baseline measurements, participants consumed 75 g glucose dissolved in two cups of non-fat milk within five minutes.
  Glucose with Whole Fat Milk: Following baseline measurements, participants consumed 75 g glucose dissolved in two cups of whole fat milk within five minutes.
  Glucose: Following baseline measurements, participants consumed a 75 g glucose solution within five minutes.
- Glucose +Non-fat Milk, Then Glucose, Then Glucose + Whole Milk: Each study day lasted approximately three hours and was separated from the other arms by four days for men and one month for women.
  Glucose with Non-fat Milk: Following baseline measurements, participants consumed 75 g glucose dissolved in two cups of non-fat milk within five minutes.
  Glucose: Following baseline measurements, participants consumed a 75 g glucose solution within five minutes.
  Glucose with Whole Fat Milk: Following baseline measurements, participants consumed 75 g glucose dissolved in two cups of whole fat milk within five minutes.
- Glucose + Whole Milk, Then Glucose, Then Glucose +Non-fat Milk: Each study day lasted approximately three hours and was separated from the other arms by four days for men and one month for women.
  Glucose with Whole Fat Milk: Following baseline measurements, participants consumed 75 g glucose dissolved in two cups of whole fat milk within five minutes.
  Glucose: Following baseline measurements, participants consumed a 75 g glucose solution within five minutes.
  Glucose with Non-fat Milk: Following baseline measurements, participants consumed 75 g glucose dissolved in two cups of non-fat milk within five minutes.
- Glucose + Whole Milk, Then Glucose +Non-fat Milk, Then Glucose: Each study day lasted approximately three hours and was separated from the other arms by four days for men and one month for women.
  Glucose with Whole Fat Milk: Following baseline measurements, participants consumed 75 g glucose dissolved in two cups of whole fat milk within five minutes.
  Glucose with Non-fat Milk: Following baseline measurements, participants consumed 75 g glucose dissolved in two cups of non-fat milk within five minutes.
  Glucose: Following baseline measurements, participants consumed a 75 g glucose solution within five minutes.
Period: Overall Study
Arm/Group | Glucose, Then Glucose +Non-fat Milk, Then Glucose + Whole Milk | Glucose, Then Glucose + Whole Milk, Then Glucose +Non-fat Milk | Glucose +Non-fat Milk, Then Glucose + Whole Milk, Then Glucose | Glucose +Non-fat Milk, Then Glucose, Then Glucose + Whole Milk | Glucose + Whole Milk, Then Glucose, Then Glucose +Non-fat Milk | Glucose + Whole Milk, Then Glucose +Non-fat Milk, Then Glucose
Started | 4 | 5 | 2 | 3 | 3 | 5
Completed | 4 | 5 | 2 | 3 | 3 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Participants who were randomized to receive either Glucose, Glucose + Whole Fat Milk, or Glucose + Non-fat Milk. All participants received all three treatments in a randomized order.
  Each study day lasted approximately three hours and was separated from the other arms by four days for men and one month for women.
  Glucose: Following baseline measurements, participants consumed a 75 g glucose solution within five minutes.
  Glucose + Whole Fat Milk: Following baseline measurements, participants consumed 75 g glucose dissolved in two cups of whole fat milk within five minutes.
  Glucose + Non-fat Milk: Following baseline measurements, participants consumed 75 g glucose dissolved in two cups of non-fat milk within five minutes.
Arm/Group | All Study Participants
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.7 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 22
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 31.6 (1.2)
Waist Circumference [Mean (Standard Deviation); unit: cm] | 107.7 (3.3)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 125.4 (2.3)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 82.7 (1.7)
Fasting Glucose [Mean (Standard Deviation); unit: mg/dL] | 109.8 (1.9)
Total Cholesterol [Mean (Standard Deviation); unit: mg/dL] | 177.7 (7.7)
Carotid Artery Intima Media Thickness (cIMT) (left) [Mean (Standard Deviation); unit: mm] — cIMT was assessed as a potential co-variate by measuring cIMT using ultrasonography
  mm | .59 (.01)
Carotid Artery Intima Media Thickness (cIMT) (right) [Mean (Standard Deviation); unit: mm] — cIMT was assessed as a potential co-variate by measuring cIMT using ultrasonography
  mm | .59 (.01)

OUTCOME MEASURES:

1. Primary Outcome: Vascular Endothelial Function
Description: Flow mediated dilation (FMD) evaluated on the basis as change from baseline to calculate FMD area under the curve from 0-180 min, i.e. i.e. Area Under the Curve (AUC) of change from baseline in FMD from 0 min to 180 min (i.e., AUC (FMD 0 min- 0 min, FMD 30 min-0 min, FMD 60 min-0 min, etc)
Time Frame: Area under curve of FMD for three hours (0, 30, 60, 90, 120, 150, and 180 min)
Measure: Mean (Standard Error); unit: %*min
Arm/Group | Glucose | Glucose With Whole Fat Milk | Glucose With Non-fat Milk
Number analyzed (Participants) | 22 | 22 | 22
%*min | -195.9 (35.99) | -6.181 (47.2) | -5.629 (36.92)

2. Secondary Outcome: Biomarker of Nitric Oxide Homeostasis (NOx)
Description: Biomarker of nitric oxide homeostasis is based on the assessment of total nitrite and nitrate concentrations. Changes relative to baseline were used to calculate area under the curve of total nitric oxide metabolites from 0-180 min, i.e. Area Under the Curve (AUC) of change from baseline in nitric oxide homeostasis from 0 min to 180 min (i.e., AUC (NOx 0 min- 0 min, NOx 30 min-0 min, NOx 60 min-0 min, etc)
Time Frame: Area under curve of nitrite/nitrate for three hours (0, 30, 60, 90, 120, 150, and 180 min)
Measure: Mean (Standard Error); unit: umol/L*min
Arm/Group | Glucose | Glucose With Whole Fat Milk | Glucose With Non-fat Milk
Number analyzed (Participants) | 22 | 22 | 22
umol/L*min | -2229 (343.3) | -1240 (252.7) | -1221 (228.3)

3. Secondary Outcome: Glucose
Description: Glucose concentrations evaluated on the basis as change from baseline to calculate glucose area under the curve from 0-180 min, i.e. Area Under the Curve (AUC) of change from baseline in glucose from 0 min to 180 min (i.e., AUC (glucose 0 min- 0 min, glucose 30 min-0 min, glucose 60 min-0 min, etc)
Time Frame: Area under curve of glucose for three hours (0, 30, 60, 90, 120, 150, and 180 min)
Measure: Mean (Standard Error); unit: mg/dL*min
Arm/Group | Glucose | Glucose With Whole Fat Milk | Glucose With Non-fat Milk
Number analyzed (Participants) | 22 | 22 | 22
mg/dL*min | 6259 (622.5) | 4481 (652.4) | 3408 (574.7)

4. Secondary Outcome: Oxidative Stress Biomarker (Malondialdehyde; MDA)
Description: MDA concentrations evaluated on the basis as change from baseline to calculate MDAarea under the curve from 0-180 min, i.e. Area Under the Curve (AUC) of change from baseline in MDA from 0 min to 180 min (i.e., AUC (MDA 0 min- 0 min, MDA 30 min-0 min, MDA 60 min-0 min, etc)
Time Frame: Area under curve of MDA for three hours (0, 30, 60, 90, 120, 150, 180 min)
Measure: Mean (Standard Error); unit: umol/L*min
Arm/Group | Glucose | Glucose With Whole Fat Milk | Glucose With Non-fat Milk
Number analyzed (Participants) | 22 | 22 | 22
umol/L*min | 54.9 (7.653) | 25.78 (9.505) | 31.3 (5.283)

ADVERSE EVENTS:
Time Frame: Participants were monitored for adverse events during the entirety of the study duration (~6 total weeks).
Description: Participants completed a cross-over trial that examined blood vessel function and related biomarkers in response to a single controlled meal. The risk for all-cause mortality relating to the study is perceived to be zero.
Arm/Group | Glucose, Then Glucose +Non-fat Milk, Then Glucose + Whole Milk | Glucose, Then Glucose + Whole Milk, Then Glucose +Non-fat Milk | Glucose +Non-fat Milk, Then Glucose + Whole Milk, Then Glucose | Glucose +Non-fat Milk, Then Glucose, Then Glucose + Whole Milk | Glucose + Whole Milk, Then Glucose, Then Glucose +Non-fat Milk | Glucose + Whole Milk, Then Glucose +Non-fat Milk, Then Glucose
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/5 | 0/2 | 0/3 | 0/3 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/5 | 0/2 | 0/3 | 0/3 | 0/5
Other Adverse Events (participants affected / at risk) | 0/4 | 0/5 | 0/2 | 0/3 | 0/3 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-02-25): https://cdn.clinicaltrials.gov/large-docs/10/NCT02482610/Prot_SAP_000.pdf